CLINICAL TRIAL: NCT01803100
Title: Study of the Temporal Profile and Bi-directional Transmission of Microorganisms Between Patients and Environmental Surfaces.
Brief Title: Characterizing and Comparing the Profile of Microorganisms From Specific Body Sites and Environmental Surfaces in Newly Disinfected Patient Rooms
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00036470; 203-1049 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Bacterial Infection
Keywords: Bacterial Colonization
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Swabs from nares, oropharynx, axillae, peri-rectal. Fecal specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized inpatients: Inpatients newly admitted into freshly-cleaned rooms.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this trial
  Other Names: There is no intervention in this trial

SUMMARY:
Overall Aim: To describe and to assess the change in the temporal profile and transmission of microorganisms between patients and environmental surfaces after admission into a newly disinfected room.

Study Activities: Investigators will prospectively and concurrently perform microbiological sampling of body sites (nose, throat, axillae, perineal and wounds) high touch surfaces (e.g. bedside rail, bed surface, toilet seat, IV pump and tray table) for consented adult patients admitted to freshly cleaned patient rooms. The microbiological sampling of body sites is already performed in many units of the hospital as standard of care. Infection and readmission related data from enrolled patients will be collected for upto 1 year after enrollment.

Data analysis: Standard surveillance for hospital-acquired infections will be performed by the infection control group of the hospital. The identity and the nature of micro-organisms colonizing the high touch surfaces of rooms and of patient's body sites will be determined and compared. Risks involved is no more than minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients who provide informed consent.

Exclusion Criteria:

* Pediatric patients under 18 years of age,
* Patients who cannot or do not provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from hospitalized inpatients who are admitted into freshly-cleaned patient rooms and provides consent to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in the Profile of Epidemiologically-Important Organism | Day 3, 7 and each week after enrollment

SECONDARY OUTCOMES:
Time to Change in the Profile of Epidemiologically Important Organism | Day 3, 7 and each week after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Luke Chen, MBBS MPH, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Durham Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina